CLINICAL TRIAL: NCT06741761
Title: The Safety and Feasibility of a 12-hour Time-Limited Enteral Feeding Protocol in Critically Ill Adults
Brief Title: 12-hour Time Limited Feeding in Critical Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Felicia Steger, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00161009
Record Dates: First submitted 2024-12-04; First posted 2024-12-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness
Keywords: time-restricted feeding; enteral feeding; critical illness; intermittent fasting
MeSH Terms: conditions — Critical Illness; Intermittent Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous 24 hour feeding (CONT24). (Active Comparator): 24 hour tube feeding is the standard of care. They will receive tube feeding continuously over 24 hours daily.
  Interventions: Other: Continuous 24 hour feeding (CONT24).
- 12-hour time-restricted feeding (TRF12) (Experimental): The 12-hour time-restricted feeding group will receive the same amount of nutrition in 12 hours as would be needed in 24 hours. The hourly feeding rate will double.
  Interventions: Other: 12-hour time-restricted feeding (TRF12)

INTERVENTIONS:
Other: 12-hour time-restricted feeding (TRF12) — The 12 hour feeding group will receive tube feeding only over a 12 hour period (6:00 AM to 6:00 PM feeding schedule).
  Arms: 12-hour time-restricted feeding (TRF12)
Other: Continuous 24 hour feeding (CONT24). — Patients in this control group will receive the standard of care which is tube feeding continuously over 24 hours.
  Arms: Continuous 24 hour feeding (CONT24).

SUMMARY:
This study is being done to assess the feasibility and safety of a time-restricted 12-hour enteral feeding protocol (experimental group) in comparison to a standard-of-care, 24-hour enteral feeding protocol (control group) in critically ill patients. Investigators hope to gain knowledge about how these feeding schedules affect feeding tolerance, blood sugar control, and other factors affecting critically ill adult patients.

* Investigators expect that the 12-hour feeding protocol will be tolerated similarly to the 24-hour feeding protocol and will not result in a greater number of adverse events related to feeding.
* Investigators expect that the proportion of participants in both groups receiving at least 75% of their estimated nutrition needs will be similar.

DETAILED DESCRIPTION:
Investigators will test a 12-hour time-restricted feeding (TRF12) protocol in critically ill adults and compare this to a standard-of-care, 24-hour continuous feeding (CONT24) schedule. Time-restricted feeding (TRF) is form of intermittent fasting involving eating within a consistent, shortened period each day, following by fasting for at least 12 hours daily. TRF may improve glycemic control, blood pressure, and circadian rhythms in metabolism relative to feeding over a longer period. In critically ill patients, most facilities feed enterally over 24-hours which may exacerbate sleep disturbances and post-intensive care syndrome. In addition to safety and feasibility measures, this 10-day trial will gather preliminary data regarding how these feeding protocols each affect glycemic control, sleep, and long-term effects of critical care, such as delirium.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age)
* With critical illness (hospitalized in an intensive care unit with a status of "ICU")
* Who have received orders for continuous enteral nutrition

Exclusion Criteria:

* "Comfort Measures Only" status
* Have orders to receive trickle feedings (feeding rate ≤10mL/hr)
* Recent surgical procedure on the GI tract (within previous 5 days at time of recruitment) or admission for GI bleed
* Receiving continuous sedation
* Expected to undergo a procedure requiring removal of study devices in the three days following enrollment
* History of malabsorptive bariatric surgery
* Admitted for a burn injury
* Known intolerance to feeding rates >100mL/hr
* Current diagnosis of pancreatitis, ileus or gastroparesis (only if using a gastrostomy tube)
* Requiring intermittent or continuous renal replacement therapy
* Pregnant or lactating
* On an intermittent feeding schedule
* Nutritional needs would require a rate higher than 120mL/hr on TRF12 protocol
* Lack of clearance by primary physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility | From randomization up to 10 days
  Safety will be measured by the need for pausing or discontinuing enteral feeds, gastrointestinal complications (including vomiting, abdominal distention, and diarrhea), other feeding complications (e.g., aspiration, gastric residuals), and hypoglycemic events. Feasibility is defined as the percentage of patients who received ≥75% of their prescribed nutrition goal, and the logistical feasibility of collecting study data.

SECONDARY OUTCOMES:
Glycemic control | From randomization up to 10 days
  Glycemic control will be assessed using a continuous glucose monitor to measure time-in-range (%), time-above-range, and number of hypoglycemic events.
Sleep quantity | From randomization up to 10 days
  Sleep quantity scores will be measured in hours using actigraphy and the Richards-Campbell Sleep questionnaire.
Circadian rhythm of skin surface temperature | From randomization up to 10 days
  Circadian rhythm of skin surface temperature will be measured across 24-hours and the phase and amplitude of the circadian rhythm of skin temperature will be quantified

OTHER OUTCOMES:
Mental health | From 1 month and 3 months post-discharge
  Mental health will be measured using the Personal Health Questionnaire-9 (PHQ-9). To provide a numerical score, we will assess anxiety, depression, and post-traumatic stress syndrome. The total score ranges from 0 to 27, with higher scores indicating more severe anxiety, depression and post-traumatic stress syndrome.
Cognitive health | From 1 month and 3 months post-discharge
  National Institutes of Health Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) will be used to assess depression or anxiety as a T-score two standard deviations above the mean. A higher score in each category indicates more of the concept being measured.
Impact of Health Status on Quality of life | From 1 month and 3 months post-discharge
  Investigators will use the Health-Related Quality of Life survey to provide a measure of the impact of health status on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Steger, PhD, MS, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided